CLINICAL TRIAL: NCT03394911
Title: The Nicholson Science Pheromone Trial
Brief Title: Healthy Adult Male Facial Skin Surface Lipid Pheromone p.o. to Treat Opioid Addiction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bubba Nicholson (Industry)
Collaborators: Tampa General Hospital (Other); Otrimed Clinical Research (Other)
Responsible Party: Sponsor-Investigator, Bubba Nicholson, Senior Scientist in Charge, Nicholson Science
Organization: Nicholson Science (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2017-12-28; First posted 2018-01-09 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Opioid Addiction; Opioid Abuse, Continuous Use; Opioid Use; Opioid-Related Disorders; Paternal Pheromone Deficiency; Opioid Dependence; Opioid Abuse; Opioid-use Disorder; Opioid Intoxication; Opioid Abuse, Episodic
MeSH Terms: conditions — Opioid-Related Disorders; Recurrence

STUDY DESIGN:
Intervention Model Description: Double-blind, cross-over, placebo-controlled clinical trial in hospital setting overseen by attending physician, χ2 test for categorized data
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical packaging, identical labeling, identifying random numbers in key onsite with pharmaceuticals technician on site. Identical vehicle. Pheromone is odorless, colorless, tasteless. Placebo handled exactly as Pheromone/experimental, but without application of pheromone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Group (Experimental): 250mg p.o. of healthy adult male facial skin surface lipid liquid pheromone on fresh, new, just-purchased, un-chewed Wrigley's Rain #5 sugarless chewing gum vehicle. 15 pieces or divided as tolerated.
  Interventions: Biological: 250mg healthy adult male facial skin surface lipid liquid pheromone
- Placebo Group (Placebo Comparator): Placebo identical to Experimental dose with randomly assigned identification numbers on unopened, unsealed key. Placebo and Experimental doses kept together and undifferentiable without the key being opened. Key available for opening 24/7 w/pharmaceuticals tech onsite. Keep pheromone/placebo doses under a fume hood. Wear 3M Versaflo activated charcoal filter supplied air respirator or equivalent to access.
  Interventions: Biological: 250mg healthy adult male facial skin surface lipid liquid pheromone

INTERVENTIONS:
Biological: 250mg healthy adult male facial skin surface lipid liquid pheromone — Human Pheromone provided p.o. to tox-screen verified opioid drug addict
  Other Names: Paternal Facial Pheromone

SUMMARY:
Healthy adult human male facial skin surface lipid liquid pheromone given by mouth to opioid addicts cures them without any withdrawal symptoms whatsoever 250mg on chewing gum vehicle by mouth. Elevated mood eventually becomes accommodated after a few weeks. The pheromone contains volatile airborne sub-pheromones which cause aversive behavior (distrust, superstition, suspicion, arrogance, astonishment/stupidity, jealousy). Artificial jealousy can be avoided by patient isolation for 40 days until the pheromone "taste" wears off the saliva. The pheromone provided is odorless, colorless, and tasteless to the conscious brain.

DETAILED DESCRIPTION:
Healthy adult human male facial skin surface lipid liquid pheromone given by mouth to opioid addicts cures them without any withdrawal symptoms whatsoever 250mg on chewing gum vehicle by mouth. Elevated mood eventually becomes accommodated after a few weeks. The pheromone contains volatile aversive sub-pheromones which cause aversive behavior (distrust, superstition, suspicion, arrogance, astonishment/stupidity, jealousy). Artificial jealousy can be avoided by patient isolation for 40 days until the pheromone "taste" wears off the saliva. The pheromone provided is odorless, colorless, and tasteless to the conscious brain. Pheromone action is insidious. The lifting of the appetite for addictive drugs "monkey on the back" feeling is gratifying. Ambition returns and ambitions are realized.

To mitigate aversive airborne sub-pheromone methyl esters (almost certainly the cause of artificial aversive emotions), we will be trying several attenuation strategies. Staff collecting, storing, and dispensing pheromone (and placebo) will utilize the provided 3M Versaflo supplied air carbon filtered respirator for pharmaceutical applications. Collection from volunteer pheromone donors and administration to tox screened opioid addicts will be in areas ventilated by Dyson carbon-filtered oscillating fans placed to break up plumes of airborne sub-pheromone sufficiently to attenuate aversive emotion. Other lab techniques will also be tried as artificially stimulated emotional and heartfelt complaints are expected, from everybody. Unfortunately, the rapid process of healing opioid addiction will involve the unavoidable creation of potentially problematic emotions. We will try smaller daily doses, reverse Fisher esterification with apple cider vinegar, more vigorous air disturbances, negative air pressure, fume hoods, isolation, etc.

ELIGIBILITY:
Inclusion Criteria: Dirty Tox Screen showing recent and continuing opioid drug dependence -

Exclusion Criteria: Pregnant people, people who desire to retain their paraphilia

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Clean Tox Screen, UDS, urinary drug screen | six weeks, all common opioids clear in six weeks time. Cannabis may take a little longer than six weeks to clear, but we are not really interested in that, are we?
  no drug use since pheromone provided. Urinary Drug Screens are among the most common medical tests in hospitals. Positive or "Dirty" urinary drug screens are routinely followed up with gas chromatography--mass spectrometry to assure test results.
Dirty Tox Screen | six weeks, all common opioids clear in six weeks time. Cannabis may take a little longer than six weeks to clear, but we are not really interested in that, are we?
  Continued heavy drug use comparable to initial Tox Screen testing. Urinary Drug Screens are among the most common medical tests in hospitals. Positive or "Dirty" urinary drug screens are routinely followed up with gas chromatography--mass spectrometry to assure test results.

CONTACTS AND LOCATIONS:
Overall Officials: Ross C Nicholson, BsIMGT, Principal Investigator — Nicholson Science

IPD SHARING:
Plan to Share IPD: Yes
Official investigations of local, state, and federal government Individual participants will be identifiable only by a random number with no identifying information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: upon publication
Access Criteria: Previously published article in med-line accessed medical journal

REFERENCES:
- [Background] Nicholson B. Does kissing aid human bonding by semiochemical addiction? Br J Dermatol. 1984 Nov;111(5):623-7. doi: 10.1111/j.1365-2133.1984.tb06635.x. No abstract available. PMID 6541944
- [Background] Nicholson B. Pheromones cause disease: pheromone/odourant transduction. Med Hypotheses. 2001 Sep;57(3):361-77. doi: 10.1054/mehy.2001.1357. PMID 11516230
- [Background] Nicholson B. Pheromones cause disease: the exocrinology of anorexia nervosa. Med Hypotheses. 2000 Mar;54(3):438-43. doi: 10.1054/mehy.1999.0872. PMID 10783484
- [Background] Nicolaides N. Skin lipids: their biochemical uniqueness. Science. 1974 Oct 4;186(4158):19-26. doi: 10.1126/science.186.4158.19. PMID 4607408